CLINICAL TRIAL: NCT00383136
Title: FATA: Comparison Between Tirofiban and Abciximab in Facilitated Angioplasty With Stent Implantation: Randomized Multicentre Study
Brief Title: FATA: Randomized Study on Facilitated Angioplasty With Tirofiban or Abciximab
Acronym: FATA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Bologna (Other)
Responsible Party: Antonio Marzocchi M.D., Istituto di Cardiologia, University of Bologna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FATA
Record Dates: First submitted 2006-09-29; First posted 2006-10-02 (Estimated); Last update posted 2008-01-16 (Estimated); Status verified 2008-01

CONDITIONS: Acute Myocardial Infarction
Keywords: STEMI; Primary Angioplasty; Abciximab; Tirofiban
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Tirofiban; Abciximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Tirofiban
  Interventions: Drug: tirofiban high-bolus dose regimen
- 2 (Active Comparator): Abciximab
  Interventions: Drug: Abciximab

INTERVENTIONS:
Drug: tirofiban high-bolus dose regimen — bolus of 25 mcg/kg of body weight, followed by 18 hours infusion of 0.15 mcg/kg/min.
  Other Names: Aggrastat
  Arms: 1
Drug: Abciximab — bolus of 0.25 mg/kg of body weight, followed by 12 hours infusion of 0.125 mcg/kg per minute
  Other Names: Reopro
  Arms: 2

SUMMARY:
The elective("standard of care") treatment of ST - elevation acute myocardial infarction (STEMI) currently consists of primary angioplasty with stent implantation during administration of Abciximab, a inhibitor of GP IIb/IIIa platelet receptor.

Tirofiban is another potent inhibitor of GP IIb/IIIa platelet receptor with an efficacy on platelet aggregation inhibition equal to or greater than Abciximab if a high dose bolus is used, i.e. 25 microg/kg, (platelet aggregation inhibition > 90% 15 minutes after infusion). It can therefore be hypothesized that this drug can improve the results of primary angioplasty to the same extent as Abciximab.

The aim of this study is to compare the efficacy, in terms of myocardial reperfusion indices, of Abciximab and high dose of Tirofiban in primary angioplasty for STEMI, both in the case of treatment before transfer and of treatment in the catheterization laboratory during the procedure.

The reference hypothesis for the study objective is the equivalence or the non-inferiority of Tirofiban with respect to Abciximab.

DETAILED DESCRIPTION:
The Facilitated Angioplasty with Tirofiban or Abciximab Study (FATA Study) is a prospective multicentre study, randomized in 2 groups (high dose Tirofiban or Abciximab), on a sample of 700 patients with acute myocardial infarction for whom primary angioplasty is indicated. Patients will be enrolled in the Emergency Room or in the Intensive Care Unit and other hospital departments or externally in the event of intervention by the Emergency Ambulance Service 118. For all these patients it must be possible to administer a IIb/IIIa inhibitor immediately after ECG and clinical diagnosis, before transfer to the cath lab for the primary angioplasty procedure. Patients arriving directly in the cath lab without being randomized before transfer will also be included.

Major exclusion criteria are: Complete left bundle branch block, Previous myocardial infarction at the same site, Post-anoxic coma, Known thrombocytopenia or leucopenia, Previous episodes of hemorrhagic diathesis or allergy to ASA or thienopyridine; Anticoagulant therapy with dicumarol with INR > 2; Previous treatment with thrombolytics (within the previous 48 hours).

Randomization will take place as soon as possible after the diagnostic ECG and will be performed by means of a centralized automatic system using SMS messages sent by ordinary cell phones.

The primary endpoint is ST resolution 90 minutes after opening of the affected vessel. Secondary endpoints include: Patency of the vessel at the first selective angiography, no reflow phenomenon during the procedure, TIMI 3 flow at the end of the procedure, MACE (death, reinfarction*, urgent TVR°) at 30 days, MACE (death, reinfarction*, TVR°) at 6 months, major bleeding requiring transfusion or surgery, or a reduction in Hb of more than 5 g%, Ictus and intracranial hemorrhage.

To demonstrate the study hypothesis, i.e. that Tirofiban is equivalent to Abciximab in facilitating primary angioplasty in acute myocardial infarction, with sufficient statistical significance, the necessary number of patients for each drug was calculated on the basis of the methods used in equivalence studies and was fixed in 350 pts per group.

390 patients have been randomized (as of Sept 15th, 2006). Results are expected by the end of 2007.

This study will establish whether in primary angioplasty a high dose of Tirofiban has an equivalent effect to Abciximab, first in terms of microcirculation protection and then of long-term clinical results. If this hypothesis is confirmed, Tirofiban could be used as an alternative to Abciximab, with considerable savings given its much lower cost.

ELIGIBILITY:
Inclusion Criteria:

1. STEMI diagnosed due to the presence of chest pain lasting at least 20 minutes and less than 6 hours, associated with elevation of the ST segment >1 mm in at least 2 adjacent leads
2. Informed consent
3. Age > 18 years

Exclusion Criteria:

1. Complete left bundle branch block
2. Previous myocardial infarction at the same site
3. Post-anoxic coma
4. Known thrombocytopenia or leucopenia
5. Severe hepatic dysfunction;
6. Previous episodes of hemorrhagic diathesis or allergy to ASA or thienopyridine;
7. Recent major surgery (< 3 months before)
8. Associated diseases that involve short life expectancy (< 2 years);
9. Arterial hypertension (AP >180/110);
10. Positive case history for stroke within the previous 30 days;
11. Positive case history for intracranial disease (aneurysm, arterovenous malformation);
12. Major trauma within the previous six weeks;
13. A clinical condition which, in the doctor's opinion, could interfere with the patient's full participation in the study;
14. Pregnancy or fertile age;
15. Anticoagulant therapy with dicumarol with INR > 2;
16. Renal insufficiency (creatinine > 3.0 mg/dl) known at the time of the study;
17. Previous treatment with thrombolytics (within the previous 48 hours);
18. Participation in other studies in progress.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 692 (Actual)
Dates: Start 2003-06; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
ST resolution | 90 minutes after opening of the IRA

SECONDARY OUTCOMES:
Patency of the IRA | at the first selective angiography
No reflow | during the procedure
TIMI 3 flow | at the end of the procedure
Myocardial blush grade | at the end of the procedure
Contractile recovery assessed with total FE and WMSI measured by echocardiography | at 48 hours and 30 days
MACE (death, reinfarction*, urgent TVR) | at 30 days
MACE (death, reinfarction*, TVR) | One year
Major bleeding requiring transfusion or surgery, or a reduction in Hb of more than 5 g%. | in-hospital
Intracranial hemorrhage. | in-hospital
Symptoms associated with new ECG alterations and a new increase in myocardial enzymes | in-hospital
Need for a new PTCA or CABG | In-hospital, 30 days, one year

CONTACTS AND LOCATIONS:
Overall Officials: ANTONIO MARZOCCHI, MD, Principal Investigator — ISTITUTO DI CARDIOLOGIA, AZIENDA OSPEDALIERA S.ORSOLA-MALPIGHI, BOLOGNA
Locations (6):
- Italy (6):
  - Divisione Di Cardiologia, Ospedale Maggiore, Bologna, BO
  - Laboratorio Di Emodinamica, Istituto Di Cardiologia, Azienda Ospedaliera S.Orsola Malpighi, Bologna, BO
  - Azienda Ospedaliera Universitaria Policlinico, Modena, MO
  - Divisione Di Cardiologia, Ospedale S.Maria Nuova, Reggio Emilia, RE
  - Divisione Di Cardiologia, Ospedale Per Gli Infermi, Rimini, RN
  - Divisione Di Cardiologia Ii, Ospedale Policlinico Le Molinette, Torino, TO

REFERENCES:
- [Derived] Marzocchi A, Manari A, Piovaccari G, Marrozzini C, Marra S, Magnavacchi P, Sangiorgio P, Marinucci L, Taglieri N, Gordini G, Binetti N, Guiducci V, Franco N, Reggiani ML, Saia F; FATA Investigators. Randomized comparison between tirofiban and abciximab to promote complete ST-resolution in primary angioplasty: results of the facilitated angioplasty with tirofiban or abciximab (FATA) in ST-elevation myocardial infarction trial. Eur Heart J. 2008 Dec;29(24):2972-80. doi: 10.1093/eurheartj/ehn467. Epub 2008 Oct 21. PMID 18940887